CLINICAL TRIAL: NCT04384835
Title: Analysis of Sexual Bias in Type 2 Innate Lymphoid Cells (ILC2) in Asthmatic Patients: Role of Androgens
Brief Title: Analysis of Sexual Bias in Type 2 Innate Lymphoid Cells (ILC2) in Asthmatic Patients
Acronym: IL-C2
Status: Completed | Type: Observational
Sponsor: University Hospital, Toulouse (Other)
Responsible Party: Sponsor
Other Study IDs: RC31/20/0007
Record Dates: First submitted 2020-03-06; First posted 2020-05-12 (Actual); Last update posted 2023-06-01 (Actual); Status verified 2023-05

CONDITIONS: Asthma
Keywords: allergy; type 2 innate lymphoid cells
MeSH Terms: conditions — Asthma; Hypersensitivity

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Mild to moderate asthma: low or medium dose of inhaled steroids according to GINA guidelines
  Interventions: Biological: Blood sample collection (one tube)
- Severe asthma: criteria described by the ATS / ERS guidelines (for the recruitment of severe patients)
  Interventions: Biological: Blood sample collection (five tubes)

INTERVENTIONS:
Biological: Blood sample collection (one tube) — Collection of one tube of 7.5 ml blood in addition to a blood sample made in clinical practice
  Groups: Mild to moderate asthma
Biological: Blood sample collection (five tubes) — Collection of five tubes of 7.5 ml blood in addition to a blood sample made in clinical practice
  Groups: Severe asthma

SUMMARY:
Asthma is more common in females than in males but the difference has not been explained yet. Group 2 innate lymphoid cells (ILC2) have recently emerged as critical players in the initiation of allergic responses but their implications in the difference between males and females in terms of asthma prevalence has not been fully studied. The aim of this project is to compare the proportion of ILC2 in blood between males and females with asthma.

DETAILED DESCRIPTION:
Asthma is more common in males until puberty but becomes more prevalent and more severe in females after puberty suggesting a protective action of male sex hormones. ILC2 have recently emerged as critical players in the initiation of allergic responses. The present team established that androgens, signaling through the nuclear receptor 3 C4 (NR3C4) androgen receptor (AR), negatively control ILC2 at steady state and during lung inflammation. Relevant to this application, females with asthma have more circulating ILC2 than males. The present hypothesis is that harnessing AR signaling in ILC2 may provide a new therapeutic approach to down regulate tissue resident ILC2. This project will analyze the sex bias in circulating ILC2 in female and male patients with moderate to severe asthma. In females with asthma, the team will purify circulating ILC2 from peripheral blood mononuclear cells (PBMC) and expand them in vitro using cytokines and stromal cells in the presence of AR antagonist or agonist ligands. Bulk ILC2 cultures at day 7 will used to measure the expression profile of various gene, including AR.

ELIGIBILITY:
Inclusion Criteria:

* Asthma according to the criteria described by Global Initiative for Asthma (GINA) guidelines
* Severe asthma according to the criteria described by the American Thoracic Society (ATS) / European Respiratory Society (ERS) guidelines (for the recruitment of severe patients)
* Mild to moderate asthma based on low or medium dose of inhaled steroids according to GINA guidelines

Exclusion Criteria:

* Asthma exacerbations defined as oral corticosteroids related to worsening respiratory symptoms within the past 4 weeks
* Pregnant women
* Breastfeeding women
* Autoimmune diseases
* Androgen medication
* Early menopause defined as the absence of menstruation for at least 1 year
* Body mass index ≥ 30 kg/m²
* Weight <40 kg
* Oral corticotherapy for more than 3 months
* Prediction of blood volume collected (care + research)> 80 ml or> 150 ml over a period of 30 days if blood collection within the past 30 days
* known anemia with hemoglobin <10 g/dl

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — The aim of this project is to compare the proportion of type 2 innate lymphoid cells (ILC2) in blood between males and females with asthma.
Study Population: Asthma patients
Sampling Method: Non-Probability Sample
Enrollment: 34 (Actual)
Dates: Start 2021-03-08 (Actual); Primary Completion 2022-05-01 (Actual); Study Completion 2023-04-12 (Actual)

PRIMARY OUTCOMES:
Frequency of circulating ILC2 between gender with asthma. | Day 1
  Estimation of the proportion of circulating ILC2 between males and females with asthma.

SECONDARY OUTCOMES:
Frequency of circulating ILC2 according to asthma severity. | Day 1
  Estimation of the proportion of circulating ILC2 between mild to moderate asthma patients and severe asthma patients.
Comparison of the effect of (androgenic receptor) AR ligands in a culture of ILC2. | Day 1
  ILC2 purified form PBMC of asthmatic females will be expanded in vitro in the presence of AR antagonist or agonist ligands. Bulk ILC2 cultures at day 7 will used to measure the expression profile of various gene, including AR.

CONTACTS AND LOCATIONS:
Overall Officials: Laurent Guilleminault, MD, Principal Investigator — University Hospital, Toulouse
Locations (1):
- Larrey hospital, Toulouse, France

IPD SHARING:
Plan to Share IPD: No